CLINICAL TRIAL: NCT02804815
Title: A Phase III, Double-blind, Placebo-controlled, Randomised Trial Assessing the Effects of Aspirin on Disease Recurrence and Survival After Primary Therapy in Common Non Metastatic Solid Tumours
Brief Title: Add-Aspirin: A Trial Assessing the Effects of Aspirin on Disease Recurrence and Survival After Primary Therapy in Common Non Metastatic Solid Tumours
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14/0814; 2013-004398-28 (EudraCT Number); 120104 (Registry Identifier: R&D)
Record Dates: First submitted 2016-02-12; First posted 2016-06-17 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Breast Cancer; Prostate Cancer; Colorectal Cancer; Gastro-oesophageal Cancer
Keywords: Aspirin; prostate; colorectal; breast; gastro-oesophageal; recurrence
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Recurrence | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aspirin 100mg (Active Comparator): Aspirin 100mg
  Interventions: Drug: Aspirin 100mg
- Placebo 100mg (Placebo Comparator): 100mg Placebo
  Interventions: Drug: Placebo 100mg
- Aspirin 300mg (Active Comparator): Aspirin 300mg
  Interventions: Drug: Aspirin 300mg
- Placebo 300mg (Placebo Comparator): 300mg Placebo
  Interventions: Drug: Placebo 300mg

INTERVENTIONS:
Drug: Aspirin 100mg — Aspirin 100mg
  Arms: Aspirin 100mg
Drug: Aspirin 300mg — Aspirin 300mg
  Arms: Aspirin 300mg
Drug: Placebo 100mg — Placebo 100mg
  Arms: Placebo 100mg
Drug: Placebo 300mg — Placebo 300mg
  Arms: Placebo 300mg

SUMMARY:
Add-Aspirin aims to assess whether regular aspirin use after standard curative therapy can prevent recurrence and improve survival in individuals with non-metastatic common tumours. The question will be assessed in four different tumour types (breast, colorectal, gastro-oesophageal and prostate) by means of parallel cohorts within an overarching trial protocol.

Eligible participants will be randomly assigned (double-blind) to either aspirin 100mg, aspirin 300mg or a matched placebo, to be taken daily for at least 5 years. Disease recurrence and survival will be assessed, along with adherence, toxicity, and other potential effects of aspirin (eg. cardiovascular).

There is a large body of evidence indicating that aspirin has anti-cancer effects. Meta-analyses of cardiovascular trials of aspirin have shown short-term effects on cancer mortality and a decrease in risk of metastases, suggesting a role for aspirin in the treatment as well as prevention of cancer. Additionally, large observational studies of individuals taking aspirin after cancer treatment have shown improved disease-specific and overall mortality for specific tumour types.

In the treatment setting, the risks of side effects associated with aspirin are expected to be outweighed by potential benefits. However, this has not yet been assessed in a randomised trial.

As a low cost, generic and widely available drug, which is generally safe, if aspirin is shown to be effective, it could have a huge impact on cancer outcomes globally.

DETAILED DESCRIPTION:
A phase III, multi-centre, double-blind, placebo-controlled randomised trial which aims to assess whether regular aspirin use after standard therapy prevents recurrence and prolongs survival in participants with non-metastatic common solid tumours.

The trial has four parallel tumour site-specific cohorts (breast, colorectal, gastro-oesophageal and prostate cancer). An overarching protocol ensures each cohort is as comparable as possible to allow a combined analysis of overall survival as a co-primary outcome measure in addition to individual tumour site-specific analyses of disease recurrence and survival.

Participants who have undergone potentially curative treatment (surgery or other radical treatment), including any standard neo-adjuvant or adjuvant therapy for breast, colorectal, gastro-oesophageal or prostate cancer or have participated in any pre-approved trials and satisfy the eligibility criteria.

Participants will be randomly assigned to 100mg aspirin, 300mg aspirin or matched placebo. All tablets will be enteric-coated to be taken daily for at least five years. Prior to randomisation, all potential participants will take open-label 100mg aspirin daily for a run-in period of approximately 8 weeks to assess tolerability and adherence.

The trial incorporates a feasibility phase during which recruitment feasibility, treatment adherence, safety and use of the run-in period will be assessed.

ELIGIBILITY:
COMMON INCLUSION CRITERIA

* Written informed consent
* WHO performance status 0, 1 or 2
* Participants should not be and have no intention of pregnancy or breast feeding during trial treatment
* Previous or current participants of other primary treatment trials if agreed in advance between trials
* No clinical or radiological evidence of residual or distant disease

BREAST COHORT INCLUSION CRITERIA

* Men or women with histologically confirmed invasive breast cancer
* Undergone complete primary invasive tumour excision with clear margins
* Surgical staging of the axilla must have been undertaken by sentinel node biopsy, axillary sampling or dissection
* In those patients with a positive sentinel node biopsy:

  o If 1, 2 or 3 nodes are positive, subsequent management of the axilla (with surgery, radiotherapy or no further intervention) should be completed prior to registration

  o If 4 or more nodes are involved, patients must have undergone completion axillary node dissection
* Radiotherapy (RT)

  * Patients who have undergone breastconserving surgery should have received adjuvant RT
  * Patients who have undergone mastectomy should have received RT if they have more than 3 axillary lymph nodes involved
  * Patients who have undergone mastectomy and have T3 tumours and/or 1, 2 or 3 involved lymph nodes may (or not) have received radiation per institutional practice
* Final histology must fall within at least one of these 3 groups:

  * Node positive
  * Node negative with highrisk features 2 or more of:

    1. ER negative
    2. HER2 positive
    3. Grade 3
    4. Lymphovascular invasion present
    5. Age <35
    6. Oncotype Dx score of >25
* In patients who have received neoadjuvant chemotherapy, patients are eligible if they have both a hormone receptor negative/HER2 negative tumour, a HER2 positive tumour or a hormone receptor positive grade 3 tumour and did not achieve a pathological complete response with neoadjuvant systemic therapy
* Known HER2 and ER status
* Timing of entry

  o If no adjuvant chemotherapy or RT: registration within 12 wks of definitive surgery achieving clear margins

  o Following adjuvant chemotherapy/RT: registration within 8 wks of last therapy.
* Participants may receive endocrine therapy and trastuzumab. All ER positive patients should be planned to undergo at least 5 yrs of adjuvant endocrine therapy.

COLORECTAL COHORT INCLUSION CRITERIA

* Histologically confirmed stage II or III adenocarcinoma of the colon or rectum and patients who have undergone resection of liver metastases with clear margins and no residual metastatic disease
* Patients with synchronous tumours if one of the tumours is at least stage II or III
* Serum CEA ideally ≤1.5 x upper limit of normal
* Have undergone curative (R0) resection with clear margins
* Timing of entry:

  * If no adjuvant treatment: registration within 12 wks of definitive surgery achieving clear margins
  * Following adjuvant treatment: registration within 8 wks of last therapy GASTROOESOPHAGEAL COHORT INCLUSION CRITERIA
* Patients with histologically confirmed adenocarcinoma, adenosquamous carcinoma or squamous cell cancer of the oesophagus, gastrooesophageal junction or stomach
* Have undergone curative (R0) resection with clear margins or primary chemoRT given with curative intent
* Timing of entry:

  * Following surgery without adjuvant treatment: registration within 12 wks of the definitive surgery achieving clear margins
  * Following primary chemoRT or surgery with adjuvant treatment: registration within 8 wks of last therapy

PROSTATE COHORT INCLUSION CRITERIA

* Men with histologically confirmed node negative nonmetastatic adenocarcinoma of the prostate
* Have undergone curative treatment, either:

  * Radical prostatectomy
  * Radical RT
* Intermediate or high risk according to D'Amico classification Depending on the curative treatment pathway, participant must additionally satisfy the following (a) Prostatectomy patients
* Open, laparoscopic or robotic radical prostatectomy
* Men treated with immediate adjuvant RT
* Men receiving adjuvant hormone therapy planned for a maximum duration of 3 yrs
* Timing of entry:

  * If no adjuvant RT: registration within 12 wks of definitive surgery and PSA at ≥6 weeks postsurgery must be <0.1ng/ml
  * Following adjuvant RT: registration within 8 wks of delivery of final fraction of RT
  * Men treated with salvage RT following a rise in PSA
* Men randomised to RADICALSHD (ISRCTN 40814031) provided all other eligibility criteria are met (b) Radical RT patients
* Men receiving neoadjuvant and/or adjuvant hormone therapy planned for a maximum duration of 3yrs
* Timing of registration within 8wks from completion of RT (c) Salvage RT patients after previous Radical Prostatectomy
* Men treated with salvage RT following a rise in PSA
* Men receiving neoand/ or adjuvant hormone therapy planned for a maximum of 3yrs

COMMON EXCLUSION CRITERIA

• Current or previous regular use of aspirin (at any dose) or current use of another NSAID for any indication.

* A past history of adverse reaction or hypersensitivity to NSAIDs, celecoxib, aspirin or other salicylates or sulphonamides, including asthma, that is exacerbated by use of NSAIDs.
* Current use of anticoagulants.
* Current or longterm use of oral corticosteroids. The treating physician should make the clinical decision whether a patient has been exposed to longterm therapy.
* Active or previous peptic ulceration
* Previous gastrointestinal bleeding except where the cause of the bleeding has been surgically removed.
* Active or previous history of inflammatory bowel disease.
* History of moderate or severe renal impairment, with eGFR<45ml/min/1.73m2.
* Previous invasive or noninvasive malignancy except:

  - DCIS where treatment consisted of resection alone. Prostate cancer initially treated with prostatectomy and now being treated with salvage radiotherapy following a rise in PSA.

  - Cervical carcinoma in situ where treatment consisted of resection alone.
  * Basal cell carcinoma where treatment consisted of resection alone or radiotherapy.
  * Superficial bladder carcinoma where treatment consisted of resection alone.
  * Other cancers where the patient has been diseasefree for ≥15 years.
* Any other physical condition which is associated with increased risk of aspirinrelated morbidity or, in the opinion of the Investigator, makes the patient unsuitable for the trial, including but not limited to severe asthma, haemophilia and other bleeding diatheses, macular degeneration and patients with a highrisk of mortality from another cause within the trial treatment period.
* Known glucose6phosphate dehydrogenase deficiency.
* LFTs greater than 1.5x the upper limit of normal unless agreed with TMG.
* Anticipated difficulties in complying with trial treatment or followup schedules.
* <16 years old.
* Participants in other treatment trials where this has not been agreed in advance by both trial teams.

BREAST COHORT EXCLUSION CRITERIA

• Metastatic or bilateral breast cancer.

COLORECTAL COHORT EXCLUSION CRITERIA • Proven (or clinically suspected) metastatic disease (patients who have undergone resection of liver metastases with clear margins and no residual metastatic disease are eligible).

GASTROOESOPHAGEAL COHORT EXCLUSION CRITERIA

• Proven (or clinically suspected) metastatic disease.

PROSTATE COHORT EXCLUSION CRITERIA

* Biopsy proven or radiologically suspected nodal involvement, or distant metastases from prostate cancer.
* Adjuvant hormone therapy planned for >3 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2015-10; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 10 years follow up
  Overall survival of all cohorts combined
Invasive disease-free survival (IDFS) | 6 years follow up
  IDFS in the breast cancer cohort
Disease-free survival (DFS) | 6 years follow up
  DFS in the colorectal cancer cohort
Overall survival | 5 years follow up
  Overall survival in the gastro-oesophageal cancer cohort
Biochemical recurrence-free survival (bRFS) | 5 years follow up
  bRFS in the prostate cancer cohort

SECONDARY OUTCOMES:
Adherence | 5 years follow up
  Patient-reported compliance (via diary card) will be assessed during the run-in period
Number of participants with serious haemorrhage (grade 3 or above) as measured by CTCAE V4.0. Data will be collected on case report forms. | 5 years follow up
Number of participants with treatment-related (active drug and placebo) cardiovascular events as assessed by CTCAE v4.0 | 5 years follow up
Number of participants with second malignancies as assessed by case report form | 5 years follow up
Number of participants that show a decline in cognition and extent of decline as assessed by the Montreal Cognitive Assessment (MoCA) | 5 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Langley, Study Director — MRC CTU at UCL
Locations (82):
- Ireland (12):
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St Luke's Hospital, Dublin
  - St Vincent's Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - University College Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - Sligo University Hospital, Sligo
  - University Hospital Waterford, Waterford
- United Kingdom (70):
  - William Harvey Hospital, Ashford
  - Stoke Mandeville Hospital, Aylesbury
  - Ysbyty Gwynedd, Bangor
  - North Devon District Hospital, Barnstaple
  - Basildon Hospital, Basildon
  - Bedford Hospital, Bedford
  - Victoria Hospital, Blackpool
  - Glan Clwyd Hospital, Bodelwyddan
  - Pilgrim Hospital, Boston
  - Royal Sussex County Hospital, Brighton
  - Bristol Haematology & Oncology Centre, Bristol
  - Fairfield Hospital, Bury
  - West Suffolk Hospital, Bury St Edmunds
  - Kent and Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - Velindre Hospital, Cardiff
  - Cumberland Infirmary, Carlisle
  - Cheltenham General Hospital, Cheltenham
  - University Hospital Coventry and Warwickshire, Coventry
  - Darlington Memorial Hospital, Darlington
  - Darent Valley Hospital, Dartford
  - Western General Hospital, Edinburgh
  - North Middlesex Hospital, Edmonton
  - Royal Devon and Exeter Hospital, Exeter
  - Queen Elizabeth Hospital, Gateshead
  - The New Victoria Hospital, Glasgow
  - Inverclyde Royal Hospital,, Greenock
  - Princess Alexandra Hospital, Harlow
  - Northwick Park Hospital, Harrow
  - Wycombe Hospital, High Wycombe
  - Hinchingbrooke Hospital, Huntingdon
  - Raigmore Hospital, Inverness
  - Ipswich Hospital, Ipswich
  - Airedale General Hospital, Keighley
  - Kidderminster General Hospital, Kidderminster
  - Kingston Hospital, Kingston
  - Royal Lancaster Infirmary, Lancaster
  - Lincoln County Hospital, Lincoln
  - Royal Marsden Hospital, London
  - St George's Hospital, London
  - Luton & Dunstable Hospital, Luton
  - Maidstone Hospital, Maidstone
  - Christie Hospital, Manchester
  - North Manchester General Hospital, Manchester
  - Wythenshawe Hospital,, Manchester
  - Queen Elizabeth The Queen Mother Hospital, Margate
  - Milton Keynes University Hospital, Milton Keynes
  - Friarage Hospital, Northallerton
  - Northampton General Hospital, Northampton
  - George Eliot Hospital, Nuneaton
  - Royal Oldham Hospital, Oldham
  - Royal Alexandra Hospital, Paisley
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire Hospital, Reading
  - Alexandra Hospital, Redditch
  - East Surrey Hospital, Redhill
  - Queen's Hospital, Romford
  - Salisbury District Hospital, Salisbury
  - Weston Park Hospital, Sheffield
  - Lister Hospital, Stevenage
  - Royal Marsden, Sutton
  - King's Mill Hospital, Sutton in Ashfield
  - Singleton Hospital, Swansea
  - Great Western Hospital, Swindon
  - Royal Cornwall Hospital, Truro
  - Weston General Hospital, Weston-super-Mare
  - West Cumberland Hospital, Whitehaven
  - Royal Albert Edward Infirmary, Wigan
  - Worcestershire Royal Hospital, Worcester
  - Wrexham Maelor Hospital, Wrexham